CLINICAL TRIAL: NCT06195670
Title: An Open-label, Multi-centered, Two-stage Clinical Study of Short-course Radiotherapy Followed by Fruquintinib Plus Sintilimab vs Bevacizumab Plus Capecitabine in the First Line Treatment of Advanced mCRC Patients Unfit for Intense Therapy
Brief Title: Clinical Study of Short-course Radiotherapy Followed by Fruquintinib Plus Sintilimab vs Bevacizumab Plus Capecitabine as First Line Treatment in Advanced mCRC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C124
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: CRC; Metastatic Colorectal Cancer; Metastatic Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; sintilimab; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCRT + fruquintinib + sintilimab (Experimental)
  Interventions: Drug: Experimental
- Bevacizumab + Capecitabine (Active Comparator)
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: Experimental — SCRT: 5*5Gy for 5 days, after a one-week rest, with fruquintinib plus sintilimab followed; Fruquintinib: qd po, 4mg/d, 2weeks on/1 week off, q3w; Sintilimab: intravenous infusion, 200mg, on day 1, q3w.
  Other Names: SCRT + fruquintinib + sintilimab
  Arms: SCRT + fruquintinib + sintilimab
Drug: Active Comparator — Capecitabine: bid po, 1000mg/m², on days 1-14, q3w; Bevacizumab: intravenous infusion, 7.5mg/kg, on day 1, q3w.
  Other Names: Bevacizumab + Capecitabine
  Arms: Bevacizumab + Capecitabine

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of short course radiotherapy followed by fruquintinib combined with Sintilimab as the first-line treatment of advanced mCRC compared to bevacizumab combined with capecitabine in patients unfit for intensive therapy.

DETAILED DESCRIPTION:
Anti-angiogenic therapy combined with immune checkpoint inhibitors in advanced mCRC has shown promising efficacy with acceptable toxicities. Radiotherapy may reshape the tumor immune microenvironment, thereby improving the efficacy of subsequent anti angiogenic drugs combined with immunotherapy.

The study is a prospective, multi-centered, two-stage clinical study with 220 unresectable advanced mCRC patients unfit for oxaliplatin or irinotecan-based intensive chemotherapy enrolled. In phase 1b, 20 patients will be recruited and the efficacy and safety of SCRT followed by fruquintinib plus sintilimab will be explored. In phase 2, 200 patients will be randomized and the efficacy and safety will be compared between SCRT followed by fruquintinib plus sintilimab and capecitabine plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent;
* 18 to 85 years old (including 18 and 85 years old);
* Histopathologically confirmed unresectable advanced metastatic colorectal adenocarcinoma;
* Have not received anti-tumor treatment for metastatic disease;
* Inability to tolerate intensive treatment regimens based on oxaliplatin or irinotecan as determined by researchers;
* At least one measurable lesion;
* Expected life expectancy ≥ 12 weeks;
* The function of important organs within the 14 days prior to enrollment meets the following requirements (no blood components or cell growth factors are allowed to be used within the 14 days prior to enrollment):
* Neutrophil absolute count ≥ 1.5 × 10^9/L;
* Platelets ≥ 80 × 10^9/L;
* Hemoglobin ≥ 8g/dL;
* Total bilirubin<1.5 times ULN;
* ALT and AST<2.5 times ULN (liver metastasis patients<5 times ULN);
* Serum creatinine ≤ 1.5 times ULN;
* Endogenous creatinine clearance rate>50ml/min;
* International standardized ratio (INR) of coagulation function ≤ 1.5 × ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
* Women of childbearing age or men whose partners have a desire to conceive should take effective contraceptive measures.

Exclusion Criteria:

* Currently has a disease or condition that affects drug absorption, or the patient is unable to take oral drugs;
* Currently has digestive tract diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectable tumors, or other conditions determined by the researcher that may cause gastrointestinal bleeding or perforation;
* History of serious cardiovascular and cerebrovascular diseases;
* Other malignant tumors within the past 5 years, excluding skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
* Clinically uncontrolled active infection, such as acute pneumonia, active hepatitis B or hepatitis C (hepatitis B virus DNA ≥ 1 × 104 copies/mL or>2000 IU/ml);
* Currently has central nervous system (CNS) metastasis or has a history of unstable or clinically symptomatic brain metastasis;
* Pregnant (positive pregnancy test before medication) or breastfeeding women;
* Urine protein ≥ 2+, or 24-hour urine protein >1.0g;
* Histologically confirmed MSI-H/dMMR tumors;
* Patients deemed unsuitable by the researchers for inclusion in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - Objective Response Rate (ORR) | From randomization until disease progression (up to approximately 3-5 years)
  ORR according to RECIST v1.1, as assessed by the Investigator
Phase 2 - Progression-free Survival (PFS) | From randomization until disease progression (up to approximately 3-5 years)
  PFS according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by the Investigator

SECONDARY OUTCOMES:
Tolerability and safety of study regimens | From randomization until the end of treatment (up to approximately 3-5 years)
  Number of Participants With Treatment-emergent Adverse Events (TEAEs) according to CTCAE v5.0
Disease Control Rate (DCR) | From randomization until disease progression (up to approximately 3-5 years)
  DCR according to RECIST v1.1, as assessed by the Investigator
Overall Survival OS) | From randomization until disease progression (up to approximately 3-5 years)
  OS according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, M.D., Principal Investigator — Zhejiang Cancer Hospital; Zhong Shi, M.D., Principal Investigator — Zhejiang Cancer Hospital; Wangxia Lv, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Ji Zhu, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No